CLINICAL TRIAL: NCT01640080
Title: A Double-Blind, Double-Randomization, Placebo-Controlled Study of the Efficacy of Intravenous Esketamine in Adult Subjects With Treatment-Resistant Depression
Brief Title: A Study of the Efficacy of Intravenous Esketamine in Adult Patients With Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR100843; ESKETIVTRD2001 (Other: Janssen Research & Development, LLC); 2011-005992-17 (EudraCT Number)
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Treatment resistant depression; Depression; Esketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Esketamine (Group 1) (Experimental)
  Interventions: Drug: Esketamine
- Esketamine (Group 2) (Experimental)
  Interventions: Drug: Esketamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esketamine — Type= exact number, number= 0.20, unit= mg/kg, form= intravenous infusion, route= intravenous use. One single intravenous infusion of esketamine 0.20 mg/kg administered on Day 1 and Day 4.
  Arms: Esketamine (Group 1)
Drug: Esketamine — Type= exact number, number= 0.40, unit= mg/kg, form= intravenous infusion, route= intravenous use. One single intravenous infusion of esketamine 0.40 mg/kg administered on Day 1 and Day 4.
  Arms: Esketamine (Group 2)
Drug: Placebo — Form= intravenous infusion, route= intravenous use. One single placebo intravenous infusion administered on Day 1 and Day 4.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy of esketamine compared with placebo in improving symptoms of depression in patients with treatment resistant depression.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor patient knows the treatment that the patient receives), double-randomization (the study drug is assigned by chance), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), multiple dose titration study in adult patients with treatment resistant depression (TRD). The study will assess the efficacy of esketamine at 24 hours after dosing on Day 1, administered as a 0.40 mg/kg and 0.20 mg/kg intravenous (i.v.) infusion, compared with placebo in improving symptoms of depression in patients with TRD, using the Montgomery-Asberg Depression Rating Scale (MADRS). The study will consist of 3 phases: a screening phase of up to 2 weeks, a 7-day double-blind treatment phase (Day 1 to Day 7), and a 4-week posttreatment (follow up) phase. The interval between the first and last dose of study medication is 3 days. The total study duration for each patient will be a maximum of 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be medically stable on the basis of clinical laboratory tests
* Diagnostic for major depressive disorder (MDD) without psychotic features
* Have an inadequate response to at least 1 antidepressant in the current episode of depression and at least one other inadequate treatment response to an antidepressant either in the current episode or in a previous episode
* Women must be not pregnant; women must be postmenopausal, surgically sterile or, if heterosexually active, practicing a highly effective method of birth control during the study and for 3 months after receiving the last dose of study drug
* Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Signed informed consent document

Exclusion Criteria:

* History of, or current signs and symptoms of diseases or conditions that would make participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments
* Has uncontrolled hypertension (systolic blood pressure (SBP)> 160 mmHg or diastolic blood pressure (DBP)> 90 mmHg despite diet, exercise or a stable dose of an allowed anti-hypertensive treatment) or any past history of hypertensive crisis
* Has known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection, or have positive results at screening
* Has a primary diagnosis of current (active) generalized anxiety disorder, panic disorder, obsessive compulsive disorder, posttraumatic stress disorder, anorexia nervosa, or bulimia nervosa
* Has a history or current diagnosis of a psychotic disorder, bipolar disorder, mental retardation, or borderline personality disorders, mood disorder with postpartum onset, somatoform disorders or chronic fatigue syndrome
* Has had major surgery, (eg, requiring general or local anesthesia) within 4 weeks before screening, or will not have fully recovered from surgery, or planned surgery during the time the subject is expected to participate in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06-27 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2013-06-03 (Actual)

PRIMARY OUTCOMES:
Change from Day 1 (baseline) to Day 2 in the Montgomery Asberg Depression Rating Scale (MADRS) total score in the double-blind treatment phase | Day 1 (baseline), Day 2
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Change from Day 1 (baseline) to Day 4 in Major Depressive Disorder (MDD) symptoms using the Montgomery Asberg Depression Rating Scale (MADRS) total score in the double-blind treatment phase | Day 1 (baseline), Day 4
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change from Day 1 (baseline) to Day 35 in Major Depressive Disorder (MDD) symptoms using the Montgomery Asberg Depression Rating Scale (MADRS) total score during the posttreatment phase | Day 1 (baseline), Day 35
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
The number of patients who have a reduction in Montgomery Asberg Depression Rating Scale (MADRS) total score of >50% versus baseline on Day 2 | Day 1 (baseline), Day 2
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change from Day 1 (baseline) to Day 4 in Major Depressive Disorder (MDD) symptoms using the Quick Inventory of Depressive Symptomatology-Self Report- 14-Item (QIDS-SR14) | Day 1 (baseline), Day 4
  The QIDS-SR14, s a version of the QIDS-SR16 with a shorter, 24-hour recall period that has been developed for this trial. The total score ranges from 0 to 27. Using a scale of severity of depression of none, mild, moderate, severe, and very severe, corresponding QIDS-SR16 total scores are none 1-5, mild 6-10, moderate 11-15, severe 16-20 and very severe 21-27.
Change from Day 1 (baseline) to Day 14 in Major Depressive Disorder (MDD) symptoms using the Quick Inventory of Depressive Symptomatology-Self Report-16-item (QIDS-SR16) | Day 1 (baseline), Day 14
  The QIDS-SR16 is a patient reported measure designed to assess the severity of depressive symptoms. The total score ranges from 0 to 27. Using a scale of severity of depression of none, mild, moderate, severe, and very severe, corresponding QIDS-SR16 total scores are none 1-5, mild 6-10, moderate 11-15, severe 16-20 and very severe 21-27.
Change from Day 1 (baseline) to Day 7 in severity of illness using the Clinical Global Impression- Severity (CGI-S) for esketamine compared to placebo | Day 1 (baseline), Day 7
  The CGI-S is a physician-rated scale that is designed to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis and improvement with treatment. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating according to: 0= not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Change from Day 1 (baseline) to Day 7 of global change in Major Depressive Disorder (MDD) since start of study treatment, as measured by the Clinical Global Impression- Improvement (CGI-I) | Day 1 (baseline), Day 7
  The CGI-I is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 0= not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Change from Day 1 (baseline) to Day 7 in severity of illness using the Patient Global Impression - Severity (PGI-S) for esketamine compared to placebo | Day 1 (baseline), Day 7
  The PGI-S is a 4-point scale that requires the patient to rate the severity of their illness at the time of assessment, relative to the patient's past experience. Considering their total experience, the patient assesses the severity of their depression illness at the time of rating as none, mild, moderate or severe.
Change from Day 1 (baseline) to Day 7 in patient perspective of global change in Major Depressive Disorder (MDD) since start of study treatment, as measured by the Patient Global Impression of Change (PGI-C) | Day 1 (baseline), Day 7
  The PGI-C is a 7-point scale that requires the patient to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the intervention. The response options are: very much improved; much improved; improved (just enough to make a difference); no change; worse (just enough to make a difference); much worse; or very much worse.
Change from Day 4 to Day 7 in Major Depressive Disorder (MDD) symptoms using the Montgomery Asberg Depression Rating Scale (MADRS) total score in the double-blind treatment phase | Day 4, Day 7
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
The number of patients who have a reduction in Montgomery Asberg Depression Rating Scale (MADRS) total score of >50% versus baseline on Day 3 | Day 1 (baseline), Day 3
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
The number of patients who have a reduction in Montgomery Asberg Depression Rating Scale (MADRS) total score of >50% versus baseline on Day 4 | Day 1 (baseline), Day 4
  The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change from Day 4 to Day 7 in Major Depressive Disorder (MDD) symptoms using the Quick Inventory of Depressive Symptomatology-Self Report- 14-Item (QIDS-SR14) | Day 4, Day 7
  The QIDS-SR14, s a version of the QIDS-SR16 with a shorter, 24-hour recall period that has been developed for this trial. The total score ranges from 0 to 27. Using a scale of severity of depression of none, mild, moderate, severe, and very severe, corresponding QIDS-SR16 total scores are none 1-5, mild 6-10, moderate 11-15, severe 16-20 and very severe 21-27.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- Belgium (4):
  - Dave
  - Ghent
  - Kortenberg
  - Lede
- Germany (4):
  - Berlin
  - Freiburg im Breisgau
  - Mainz
  - München
- Gdansk, Poland

REFERENCES:
- [Derived] Lewis S, Romano C, De Bruecker G, Murrough JW, Shelton R, Singh JB, Jamieson C. Analysis of Clinical Trial Exit Interview Data in Patients with Treatment-Resistant Depression. Patient. 2019 Oct;12(5):527-537. doi: 10.1007/s40271-019-00369-8. PMID 31270774
- [Derived] Johnson KM, Devine JM, Ho KF, Howard KA, Saretsky TL, Jamieson CA. Evidence to Support Montgomery-Asberg Depression Rating Scale Administration Every 24 Hours to Assess Rapid Onset of Treatment Response. J Clin Psychiatry. 2016 Dec;77(12):1681-1686. doi: 10.4088/JCP.15m10253. PMID 28086004
- [Derived] Singh JB, Fedgchin M, Daly E, Xi L, Melman C, De Bruecker G, Tadic A, Sienaert P, Wiegand F, Manji H, Drevets WC, Van Nueten L. Intravenous Esketamine in Adult Treatment-Resistant Depression: A Double-Blind, Double-Randomization, Placebo-Controlled Study. Biol Psychiatry. 2016 Sep 15;80(6):424-431. doi: 10.1016/j.biopsych.2015.10.018. Epub 2015 Nov 3. PMID 26707087